CLINICAL TRIAL: NCT07320482
Title: A Retrospective Observational Study Evaluating Surgical Strategies and Safety Profiles of Cochlear Implantation in Pediatric Patients With CHARGE Syndrome
Brief Title: A Strategic Approach to Safe and Effective Cochlear Implantation in Patients With CHARGE Syndrome
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Choi Byung Yoon, Professor of Otolaryngology-Head and Neck Surgery Investigator Affiliation: Seoul National University Bundang Hospital, Seoul National University Bundang Hospital
Other Study IDs: B-2512-1012-104
Record Dates: First submitted 2025-11-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: CHARGE Syndrome
MeSH Terms: conditions — CHARGE Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (Observation Study)

SUMMARY:
This retrospective observational study aims to evaluate cochlear anatomy, surgical challenges, and strategic approaches for safe cochlear implantation in pediatric patients with CHARGE syndrome. CHARGE syndrome is frequently associated with complex temporal bone malformations, which may increase the risk of intraoperative complications and limit the applicability of standard surgical techniques.

The investigators reviewed preoperative imaging findings, operative records, and perioperative clinical data from pediatric patients with CHARGE syndrome who underwent cochlear implantation at Seoul National University Bundang Hospital. The objective of this study is to identify anatomical variations, characterize surgical difficulties, and describe practical surgical strategies that may enhance safety during cochlear implantation in this high-risk population.

The findings of this study are expected to contribute to improved understanding of cochlear and temporal bone anatomy in CHARGE syndrome and to support safer and more effective surgical planning for affected pediatric patients.

DETAILED DESCRIPTION:
This retrospective observational study evaluates surgical strategies and safety profiles of cochlear implantation in pediatric patients diagnosed with CHARGE syndrome. Medical records, preoperative imaging studies (CT and/or MRI), and operative reports were retrospectively reviewed to assess cochlear and temporal bone anatomy, surgical challenges, and intraoperative findings.

The study focuses on identifying anatomical variations commonly encountered in CHARGE syndrome and describing practical surgical approaches used to manage complex inner ear and temporal bone malformations. No interventions were assigned as part of this observational study.

ELIGIBILITY:
* Inclusion Criteria

  * Pediatric patients diagnosed with CHARGE syndrome
  * Underwent cochlear implantation at Seoul National University Bundang hospital
  * Availability of preoperative imaging (CT and/or MRI)
  * Complete operative records available
* Exclusion Criteria -Patients with CHARGE syndrome who did not undergo cochlear implantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of pediatric patients diagnosed with CHARGE syndrome who underwent cochlear implantation at Seoul National University Bundang Hospital. These patients typically present with complex inner ear and temporal bone malformations, including cochlear hypoplasia, semicircular canal anomalies, and aberrant facial nerve courses. All participants included in this retrospective review had available preoperative imaging (CT and/or MRI) and complete operative records.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2025-11-21 (Actual); Primary Completion 2025-11-22 (Actual); Study Completion 2025-11-22 (Actual)

PRIMARY OUTCOMES:
"Characterization of Cochlear and Temporal Bone Anatomical Abnormalities in Pediatric Patients With CHARGE Syndrome" | Preoperative (Baseline)
  This outcome evaluates the type and severity of cochlear, vestibular, and temporal bone malformations based on retrospective review of preoperative radiologic imaging, including computed tomography (CT) and magnetic resonance imaging (MRI), as documented in existing medical records.
"Characterization of Cochlear and Temporal Bone Anatomical Abnormalities in Pediatric Patients With CHARGE Syndrome" | Preoperative (Baseline)
  From existing medical records and preoperative imaging (CT/MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Kyeonggido, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study involves a small cohort of pediatric patients with CHARGE syndrome, a rare condition in which the risk of re-identification is high even after de-identification. The dataset includes sensitive clinical details, imaging findings, and operative records that cannot be safely disclosed under institutional privacy and ethical policies